CLINICAL TRIAL: NCT07215910
Title: Phase III Trial of Radiotherapy Followed by Adjuvant Temozolomide in Combination With the IDH Inhibitor Vorasidenib vs Placebo in IDH-Mutated Newly-Diagnosed Grade 3 Astrocytomas
Brief Title: Testing Addition of an Anti-cancer Drug, Vorasidenib to Temozolomide, After Radiation for Advanced Brain Cancer
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A072301
Record Dates: First submitted 2025-10-09; First posted 2025-10-14 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Astrocytoma, IDH-Mutant, Grade 3
MeSH Terms: conditions — Astrocytoma; Lymphoma, Follicular | interventions — Radiotherapy, Intensity-Modulated; Temozolomide; vorasidenib; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (temozolomide, placebo) (Placebo Comparator): Patients receive IMRT/VMAT or PBS or IMPT QD on Monday-Friday for 33 fractions. Starting 4 weeks after radiotherapy, patients receive temozolomide PO QD on days 1-5 and placebo PO QD on days 1-28 of each cycle. Cycles of combination treatment repeat every 28 days for up to 12 months and placebo alone repeats every 28 days in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo blood sample collection and MRI throughout the study.
  Interventions: Radiation: Intensity-Modulated Radiation Therapy; Radiation: Volume Modulated Arc Therapy; Radiation: Pencil Beam Scanning; Procedure: Intensity-Modulated Proton Therapy; Drug: Temozolomide; Drug: Placebo Administration; Procedure: Biospecimen Collection; Procedure: Magnetic Resonance Imaging; Other: Questionnaire Administration
- Arm II (temozolomide, vorasidenib) (Experimental): Patients receive IMRT/VMAT or PBS or IMPT QD on Monday-Friday for 33 fractions. Starting 4 weeks after radiotherapy, patients receive temozolomide PO QD on days 1-5 and vorasidenib PO QD on days 1-28 of each cycle. Cycles of combination treatment repeat every 28 days for up to 12 months and vorasidenib alone repeats every 28 days in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo blood sample collection and MRI throughout the study.
  Interventions: Radiation: Intensity-Modulated Radiation Therapy; Radiation: Volume Modulated Arc Therapy; Radiation: Pencil Beam Scanning; Procedure: Intensity-Modulated Proton Therapy; Drug: Temozolomide; Drug: Vorasidenib; Procedure: Biospecimen Collection; Procedure: Magnetic Resonance Imaging; Other: Questionnaire Administration

INTERVENTIONS:
Radiation: Intensity-Modulated Radiation Therapy — Undergo IMRT/VMAT
  Other Names: IMRT
Radiation: Volume Modulated Arc Therapy — Undergo IMRT/VMAT
  Other Names: VMAT
Radiation: Pencil Beam Scanning — Undergo PBS
  Other Names: PBS
Procedure: Intensity-Modulated Proton Therapy — Undergo IMPT
  Other Names: IMPT
Drug: Temozolomide — Given PO
Drug: Vorasidenib — Given PO
  Arms: Arm II (temozolomide, vorasidenib)
Drug: Placebo Administration — Given PO
  Arms: Arm I (temozolomide, placebo)
Procedure: Biospecimen Collection — Undergo blood sample collection
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: MRI
Other: Questionnaire Administration — Ancillary Studies

SUMMARY:
This phase III trial compares the effect of vorasidenib to placebo in combination with usual treatment, temozolomide, in treating patients with newly diagnosed grade 3 astrocytoma after radiation. Temozolomide is in a class of medications called alkylating agents. It works by damaging the cell's deoxyribonucleic acid and may kill tumor cells and slow down or stop tumor growth. Vorasidenib citrate blocks the proteins made by the mutated IDH1 and IDH2 genes, which may help keep tumor cells from growing. It is a type of enzyme inhibitor and a type of targeted therapy. Adding vorasidenib to the usual treatment, temozolomide, may be more effective than temozolomide alone in treating patients with newly diagnosed grade 3 astrocytoma after radiation therapy.

DETAILED DESCRIPTION:
The primary and secondary objectives of the study:

PRIMARY OBJECTIVE:

I. To determine if vorasidenib citrate (vorasidenib) and adjuvant temozolomide following radiation therapy improves progression-free survival (PFS) per blinded independent review in patients with newly-diagnosed IDH-mutant astrocytoma (World Health Organization [WHO] grade 3) compared to placebo given with adjuvant temozolomide following radiation therapy.

SECONDARY OBJECTIVES:

I. To evaluate the safety and tolerability of vorasidenib versus (vs.) placebo in combination with temozolomide, following radiation therapy.

II. To evaluate PFS associated with vorasidenib vs. placebo in combination with temozolomide following radiation therapy, defined by local institutional review.

III. To evaluate the efficacy of vorasidenib vs. placebo in combination with adjuvant temozolomide, following radiation therapy, based on overall survival (OS).

IV. To evaluate the efficacy of vorasidenib vs. placebo in combination with temozolomide, following radiation therapy, based on objective response rate (ORR), complete response (CR) + partial response (PR), time to response, time to CR+PR, duration of response, and duration of CR+PR, with response assessed per the blinded independent review using the Response Assessment in Neuro-Oncology (RANO) 2.0 criteria in patients with measurable tumor at baseline.

V. To evaluate the efficacy of vorasidenib vs. placebo in combination with temozolomide, following radiation therapy, based on ORR, CR+PR, time to response, time to CR+PR, duration of response, and duration of CR+PR, with response assessed per local institutional review or investigator using the RANO 2.0 criteria.

VI. To evaluate the efficacy of vorasidenib vs. placebo in combination with temozolomide, following radiation therapy, based on time to next intervention.

VII. To evaluate vorasidenib vs. placebo in combination with temozolomide, following radiation, with respect to health-related quality of life (HRQoL) as assessed by the Functional Assessment of Cancer Therapy-Brain (FACT-Br) and symptom burden as assessed by the MD Anderson Symptom Inventory-Brain Tumor (MDASI-BT).

EXPLORATORY OBJECTIVES:

I. To correlate tumor genotype with PFS. II. To evaluate the effect of the addition of vorasidenib to adjuvant temozolomide on seizure control.

OUTLINE: Patients are randomized 1:1 to 1 of 2 arms.

ARM I (CONTROL): Patients receive intensity-modulated radiation therapy (IMRT)/volume modulated arc therapy (VMAT) or pencil beam scanning (PBS) or intensity-modulated proton therapy (IMPT) once daily (QD) on Monday-Friday for 33 fractions. Starting 4 weeks after radiotherapy, patients receive temozolomide orally (PO) QD on days 1-5 and placebo PO QD on days 1-28 of each cycle. Cycles of combination treatment repeat every 28 days for up to 12 months and placebo alone repeats every 28 days in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo blood sample collection and magnetic resonance imaging (MRI) throughout the study.

ARM II (EXPERIMENTAL): Patients receive IMRT/VMAT or PBS or IMPT QD on Monday-Friday for 33 fractions. Starting 4 weeks after radiotherapy, patients receive temozolomide PO QD on days 1-5 and vorasidenib PO QD on days 1-28 of each cycle. Cycles of combination treatment repeat every 28 days for up to 12 months and vorasidenib alone repeats every 28 days in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo blood sample collection and MRI throughout the study.

After completion of study treatment, patients are followed up every 3 months for the first 2 years, every 4 months for the next 2 years, and then every 6 months for up to 10 years.

ELIGIBILITY:
Inclusion Criteria:

* STEP 0: Histologic diagnosis of astrocytoma, IDH-mutant (central nervous system [CNS] WHO grade 3)
* STEP 0: Available diagnostic slides (hematoxylin and eosin staining method [H&E] and immunohistochemical stains for central review)
* STEP 0: Tissue available for central biomarker testing (CDKN2A/B and1p/19q co-deletion [all patients], and IDH1/IDH2 [if needed])
* STEP 1: Centrally-confirmed diagnosis of astrocytoma, IDH-mutant (CNS WHO grade 3)
* STEP 1: Presence of IDH1 p.R132 or IDH2 p.172 mutation, confirmed by central review of immunohistochemical stain or molecular testing results, with central confirmation of equivocal results
* STEP 1: Absence of CDKN2A/B homozygous deletion by central testing
* STEP 1: Absence of whole arm 1p/19q co-deletion (i.e. intact 1p/19q) by central testing
* STEP 1: No evidence of spinal or leptomeningeal disease
* STEP 1: No prior chemotherapy, cranial irradiation, IDH-inhibitor therapy, radiotherapy, vaccine therapy, small-molecule therapy, or laser ablation
* STEP 1: Prior diagnostic surgery/resection/biopsy ≤ 6 months of registration
* STEP 1: Planned radiotherapy and adjuvant chemotherapy
* STEP 1: Age ≥ 12 years
* STEP 1: Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 (or Karnofsky performance status [KPS] ≥ 60%)
* STEP 1: Absolute neutrophil count (ANC) ≥ 1,500/mm^3
* STEP 1: Hemoglobin ≥ 9 g/dL
* STEP 1: Platelet count ≥ 100,000/mm^3
* STEP 1: Total bilirubin ≤ 1.5 x upper limit of normal (ULN)

  * For patients with Gilbert syndrome, total bilirubin ≤ 1.0 x ULN
* STEP 1: Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT)(serum glutamic pyruvic transaminase [SGPT]) ≤ 2.5 x ULN
* STEP 1: Alkaline phosphatase ≤ 2.5 x ULN
* STEP 1: Creatinine ≤ 2.0 x ULN or calculated (calc.) creatinine clearance > 40 mL/min

  * For patients ≥ 18 years of age, calculated using the Cockcroft-Gault equation. For patients < 18 years of age, calculated using the Bedside Schwartz method:
  * Age: 10 to < 13 years; Maximum Serum Creatinine (mg/dL): 1.2 (male) 1.2 (female)
  * Age: 13 to < 16 years; Maximum Serum Creatinine (mg/dL): 1.5 (male) 1.4 (female)
  * Age: ≥ 16 years; Maximum Serum Creatinine (mg/dL): 1.7(male) 1.4 (female)
* STEP 1: Not pregnant and not nursing, because this study involves agents whose genotoxic, mutagenic, and teratogenic effects on the developing fetus and newborn are unknown

  * Therefore, for women of childbearing potential only, a negative pregnancy test done ≤ 14 days prior to registration is required
* STEP 1: Women and men of reproductive potential should agree to abstain from sexual intercourse or use two highly effective methods of birth control, at least one of which must be a barrier method, throughout their participation in this study and for at least 90 days after the last dose of vorasidenib. Reproductive status and discussions about birth control measures should be documented in the patient's record. Abstinence is acceptable only as true abstinence when this is in line with the preferred and usual lifestyle of the patient; periodic abstinence (e.g. calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of birth control. Highly effective forms of birth control are defined as hormonal oral contraceptives, injectables, patches, intrauterine devices, intrauterine hormone release systems, bilateral tubal ligation, condoms with spermicide, or male partner sterilization
* STEP 1: No severe or intercurrent illness, no active infection that requires systemic anti-infective therapy, and no active infection with an unexplained fever > 38.5°C within 7 days prior to registration
* STEP 1: Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* STEP 1: Patients must be able to tolerate or undergo an MRI
* STEP 1: Patients with known HIV infection on effective anti-retroviral therapy with undetectable viral load within 6 months prior to registration are eligible for this trial
* STEP 1: For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* STEP 1: Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* STEP 1: No significant active cardiac disease within 6 months prior to registration, including New York Heart Association Functional Classification class III or IV congestive heart failure, myocardial infarction, unstable angina, and/or stroke. To be eligible for this trial, patients should be class 2B or better
* STEP 1: No history of significant (grade ≥ 2) intratumoral or peri-tumoral hemorrhage
* STEP 1: No known active inflammatory gastrointestinal disease, chronic diarrhea, prior gastric resection or lap band dysphagia, short-gut syndrome, gastroparesis, or other condition causing an inability to swallow oral formulations of agents. Gastroesophageal reflux disease under medical treatment is allowed (assuming no drug interaction potential)
* STEP 1: No known hypersensitivity to any of the components of vorasidenib or temozolomide
* STEP 1: No other acute or chronic medical condition or laboratory abnormality that may increase the risk associated with study participation or protocol therapy administration or may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the patient inappropriate for entry into this study
* STEP 1: No concurrent use of other investigational agents
* STEP 1: No concurrent use of alternating tumor treating field (TTField) therapy
* STEP 1: No concurrent use of therapeutic doses of steroids for glioma. Concurrent use of physiologic doses of steroids (defined as equivalent of ≤ 10 mg prednisone daily) for medical conditions unrelated to glioma is allowed. Corticosteroids administered for reasons related to glioma should be used in the smallest dose possible to control symptoms of cerebral edema and mass effect and discontinued whenever possible.
* STEP 1: No concurrent use of warfarin sodium or any other Coumadin-derivative anticoagulant. Patients must be off Coumadin-derivative anticoagulants for at least 7 days prior to registration. Low molecular weight heparin (LMWH) and factor Xa inhibitors are allowed
* STEP 1: No concurrent use of strong and moderate CYP1A2 inhibitors, moderate CYP1A2 inducers, or CYP3A substrates where a minimal concentration change can reduce efficacy. Patients should be transferred to other medications prior to registration

Exclusion Criteria:

-

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 408 (Estimated)
Dates: Start 2025-10-20 (Estimated); Primary Completion 2033-05-31 (Estimated); Study Completion 2040-01 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) by blinded independent central review (BICR) | assessed up to 10 years
  This is defined as the time from randomization to the time of documented disease progression, as determined by BICR using the Response Assessment in Neuro-Oncology (RANO) 2.0 criteria or death due to any cause. PFS distributions will be evaluated for each arm and will be graphically and quantitatively compared using Kaplan-Meier methods. These methods will be used to estimate the median PFS as well as 2-, 3-, and 5-year estimates for PFS by treatment arm along with corresponding 95% confidence intervals. Cox proportional hazards models will also be used to assess influential factors on PFS both in the univariate and the multivariable settings.

SECONDARY OUTCOMES:
Progression free survival (PFS) by local review | up to 10 years
  This is defined as the time from randomization to the time of documented disease progression, as determined by local (institutional/investigator) review using the Response Assessment in Neuro-Oncology (RANO) 2.0 criteria or death due to any cause. PFS distributions will be evaluated for each arm and will be graphically and quantitatively compared using Kaplan-Meier methods. These methods will be used to estimate the median PFS as well as 2-, 3-, and 5-year estimates for PFS by treatment arm along with corresponding 95% confidence intervals. Cox proportional hazards models will also be used to assess influential factors on PFS both in the univariate and the multivariable settings.
Incidence of adverse events (AEs) | Up to 30 days after last dose of study treatment
  AEs will be evaluated by treatment regimen. Will be summarized per the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0 and where toxicities will be defined as AEs that are deemed to be at least possibly treatment-related. The maximum grade for each type of treatment-related AE will be recorded for each patient, and the frequency of each will be summarized by treatment arm. Frequency tables and graphical evaluations of AEs and treatment-related AEs will be summarized and evaluated to assess if there are any patterns or differences in the rates or types of AEs.
Overall survival (OS) | up to 10 years
  This is defined as the time from randomization to the date of death due to any cause. Distributions will be evaluated for each arm using the Kaplan Meier method to calculate 2-, 3-, and 5-year rates along with corresponding 95% confidence intervals. Distributions will be compared between arms using the log rank test.
Objective response rate (ORR) by blinded independent central review (BICR) | up to 10 years
  Will be summarized by treatment arm. This is defined as the proportion of patients with measurable tumor at baseline who achieve a minor, partial, or complete response to therapy divided by the total number of patients with measurable tumor at baseline who were randomized and treated on that arm. Response will be determined by BICR using the Response Assessment in Neuro-Oncology (RANO) 2.0 criteria. Assuming the number of patients who respond to therapy on each arm is binomially distributed, these proportions along with corresponding 95% confidence intervals will be estimated.
Complete response (CR) + partial response (PR) rate by blinded independent central review (BICR) | up to 10 years
  Will be summarized by treatment arm. This is defined as the proportion of patients with measurable tumor at baseline who achieve a partial or complete response to therapy divided by the total number of patients with measurable tumor at baseline who were randomized and treated on that arm. Response will be determined by BICR using the Response Assessment in Neuro-Oncology (RANO) 2.0 criteria. Assuming the number of patients who respond to therapy on each arm is binomially distributed, these proportions along with corresponding 95% confidence intervals will be estimated.
Time to response by blinded independent central review (BICR) | up to 10 years
  Will be summarized by treatment arm. This is defined only for patients with measurable disease at baseline as the time from randomization to the date of response to treatment (minor, partial, or complete), as determined by BICR using the Response Assessment in Neuro-Oncology (RANO) 2.0 criteria. Distributions will be evaluated for each arm using the Kaplan Meier method to calculate 6- and 12-month rates along with corresponding 95% confidence intervals.
Time to complete response (CR) + partial response (PR) by blinded independent central review (BICR) | up to 10 years
  Will be summarized by treatment arm. This is defined only for patients with measurable disease at baseline as the time from randomization to the date of response to treatment (partial or complete), as determined by BICR using the Response Assessment in Neuro-Oncology (RANO) 2.0 criteria. Distributions will be evaluated for each arm using the Kaplan Meier method to calculate 6- and 12-month rates along with corresponding 95% confidence intervals.
Duration of response by blinded independent central review (BICR) | up to 10 years
  Will be summarized by treatment arm for only patients who had measurable disease at baseline and achieved a response (minor, partial, or complete) while on treatment, as determined by BICR using the Response Assessment in Neuro-Oncology (RANO) 2.0 criteria. This is defined as the time from the date of response to treatment (minor, partial, or complete) until the date of progression, as determined by BICR. Distributions will be evaluated for each arm using the Kaplan Meier method to calculate 1- and 2-year rates along with corresponding 95% confidence intervals.
Duration of Complete response (CR) + partial response (PR) by blinded independent central review (BICR) | up to 10 years
  Will be summarized by treatment arm for only patients who had measurable disease at baseline and achieved a response (partial or complete) while on treatment, as determined by BICR using the Response Assessment in Neuro-Oncology (RANO) 2.0 criteria. This is defined as the time from the date of response to treatment (partial or complete) until the date of progression, as determined by BICR. Distributions will be evaluated for each arm using the Kaplan Meier method to calculate 1- and 2-year rates along with corresponding 95% confidence intervals.
Objective response rate (ORR) by local review | up to 10 years
  Will be summarized by treatment arm. This is defined as the proportion of patients with measurable tumor at baseline who achieve a minor, partial, or complete response to therapy divided by the total number of patients with measurable tumor at baseline who were randomized and treated on that arm. Response will be determined by local, institutional / investigator review using the Response Assessment in Neuro-Oncology (RANO) 2.0 criteria. Assuming the number of patients who respond to therapy on each arm is binomially distributed, these proportions along with corresponding 95% confidence intervals will be estimated.
Complete response (CR) + partial response (PR) rate by local review | up to 10 years
  Will be summarized by treatment arm. This is defined as the proportion of patients with measurable tumor at baseline who achieve a partial or complete response to therapy divided by the total number of patients with measurable tumor at baseline who were randomized and treated on that arm. Response will be determined by local, institutional / investigator review using the Response Assessment in Neuro-Oncology (RANO) 2.0 criteria. Assuming the number of patients who respond to therapy on each arm is binomially distributed, these proportions along with corresponding 95% confidence intervals will be estimated.
Time to response by local review | up to 10 years
  Will be summarized by treatment arm. This is defined only for patients with measurable disease at baseline as the time from randomization to the date of response to treatment (minor, partial, or complete), as determined by local, institutional / investigator review using the Response Assessment in Neuro-Oncology (RANO) 2.0 criteria. Distributions will be evaluated for each arm using the Kaplan Meier method to calculate 6- and 12-month rates along with corresponding 95% confidence intervals.
Time to complete response (CR) + partial response (PR) by local review | up to 10 years
  Will be summarized by treatment arm. This is defined only for patients with measurable disease at baseline as the time from randomization to the date of response to treatment (partial or complete), as determined by local, institutional / investigator review using the Response Assessment in Neuro-Oncology (RANO) 2.0 criteria. Distributions will be evaluated for each arm using the Kaplan Meier method to calculate 6- and 12-month rates along with corresponding 95% confidence intervals.
Duration of response by local review | up to 10 years
  Will be summarized by treatment arm for only patients who had measurable disease at baseline and achieved a response (minor, partial, or complete) while on treatment, as determined by local, institutional / investigator review using the Response Assessment in Neuro-Oncology (RANO) 2.0 criteria. This is defined as the time from the date of response to treatment (minor, partial, or complete) until the date of progression, as determined by local review. Distributions will be evaluated for each arm using the Kaplan Meier method to calculate 1- and 2-year rates along with corresponding 95% confidence intervals.
Duration of Complete response (CR) + partial response (PR) by local review | up to 10 years
  Will be summarized by treatment arm for only patients who had measurable disease at baseline and achieved a response (partial or complete) while on treatment, as determined by local, institutional / investigator review using the Response Assessment in Neuro-Oncology (RANO) 2.0 criteria. This is defined as the time from the date of response to treatment (partial or complete) until the date of progression, as determined by local review. Distributions will be evaluated for each arm using the Kaplan Meier method to calculate 1- and 2-year rates along with corresponding 95% confidence intervals.
Time to next therapeutic intervention | up to 10 years
  Will be summarized by treatment arm. This is defined as the time from randomization to the time of first subsequent non-protocol treatment. Distributions will be evaluated for each arm using the Kaplan Meier method to calculate 2-, 3-, and 5-year rates along with corresponding 95% confidence intervals.

OTHER OUTCOMES:
Health related quality of life | up to 3 years
  Will be assessed using the Functional Assessment of Cancer Therapy-Brain (FACT-BR). The total score ranges from 0 to 200, with higher score indicating better quality of life.
Symptom burden | up to 3 years
  Will be assessed using the MD Anderson Symptom Inventory-Brain Tumor (MDASI-BT). It consists of 23 symptoms rated on an 11-point scale (0 to 10) to indicate the presence and severity of the symptom, with 0 being "not present" and 10 being "as bad as you can imagine.
Correlation of tumor genotype with PFS | up to 10 years
  Testing of banked biospecimens to determine tumor genotypes will not be conducted until a protocol amendment or separate correlative science proposal is approved. Details of planned statistical analyses will be included in the amendment or proposal.
Effect of the addition of vorasidenib to adjuvant temozolomide on seizure control | up to 10 years
  Results from the MD Anderson Symptom Inventory-Brain Tumor (MDASI-BT) question for severity of seizures will be compared between arms.

CONTACTS AND LOCATIONS:
Overall Officials: Ugonma N Chukwueke, MD, Study Chair — Alliance for Clinical Trials in Oncology; Rifaquat M. Rahman, MD, Study Chair — Alliance for Clinical Trials in Oncology; Patrick Y Wen, MD, Study Chair — Alliance for Clinical Trials in Oncology

IPD SHARING:
Plan to Share IPD: Undecided